CLINICAL TRIAL: NCT00232167
Title: Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Of The Efficacy And Tolerability Of Indiplon Therapy Initiated With Sertraline Versus Sertraline Monotherapy In Subjects With Insomnia And Co-Existing Major Depressive Disorder
Brief Title: Study Of Indiplon/Placebo With Sertraline In Insomnia Co-Existing With Depression
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Please see Detailed Description below for termination reason.
Sponsor: Neurocrine Biosciences (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5761022
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2007-10-02 (Estimated); Status verified 2007-10

CONDITIONS: Insomnia; Depression
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression | interventions — indiplon; Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Indiplon
Drug: Sertraline

SUMMARY:
The goal of this study is to determine whether indiplon, when administered with sertraline, improves insomnia symptoms and depressive symptoms in subjects with both insomnia and depression.

DETAILED DESCRIPTION:
This Pfizer run study stopped due to the co-development program for indiplon being terminated between Pfizer and Neurocrine. The study was terminated on 16 November 2006. There were no safety issues leading to the decision to terminate this study.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV defined insomnia
* DSM-IV defined Major Depression

Exclusion Criteria:

* Current suicidal ideation or behavior
* Primary sleep disorder other than insomnia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380
Dates: Start 2005-11; Study Completion 2006-04

PRIMARY OUTCOMES:
Change from baseline to week 1 in subjective total sleep time (sTST); (average of the week one data)

SECONDARY OUTCOMES:
Change from baseline in subjective total sleep time (sTST). Change from baseline in subjective parameters: LSO, sWASO, sNAASO, Sleep Quality (IVR). Change from baseline in the 3-item HAM-D insomnia factor (items #4-6).